CLINICAL TRIAL: NCT05282797
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Doses of CB1 Antagonist ANEB-001 in Healthy Occasional Cannabis Users in a THC Challenge Test.
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CB1 Antagonist ANEB-001 in a THC Challenge Test
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anebulo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN01AC11
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Acute Cannabinoid Intoxication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Part A - ANEB-001 (Experimental): Subjects receive THC and varying amounts of ANEB-001
  Interventions: Drug: ANEB-001
- Part A - Placebo (Placebo Comparator): Subjects receive THC and placebo
  Interventions: Drug: Placebo
- Part B - Cohort 1 - ANEB-001 (Experimental): Subjects receive 21 mg of THC and 30 mg of ANEB-001
  Interventions: Drug: ANEB-001
- Part B - Cohort 1 - Placebo (Placebo Comparator): Subjects receive 21 mg of THC and placebo
  Interventions: Drug: Placebo
- Part B - Cohort 2 - ANEB-001 (Experimental): Subjects receive 21 mg of THC and 10 mg of ANEB-001
  Interventions: Drug: ANEB-001
- Part B - Cohort 2 - Placebo (Placebo Comparator): Subjects receive 21 mg of THC and placebo
  Interventions: Drug: Placebo
- Part B - Cohort 3 - ANEB-001 (Experimental): Subjects receive 21 mg of THC and 1 hour later, 30 mg ANEB-001
  Interventions: Drug: ANEB-001
- Part B - Cohort 3 - Placebo (Placebo Comparator): Subjects receive 21 mg THC and 1 hour later, placebo
  Interventions: Drug: Placebo
- Part B - Cohort 4 - ANEB-001 (Experimental): Subjects receive 40 mg of THC and 1 hour later, 10 mg of ANEB-001
  Interventions: Drug: ANEB-001
- Part B - Cohort 4 - Placebo (Placebo Comparator): Subjects receive 40 mg of THC and 1 hour later, placebo
  Interventions: Drug: Placebo
- Part B - Cohort 5 - ANEB-001 (Experimental): Subjects receive 30 mg of THC and 1 hour later, 10 mg of ANEB-001
  Interventions: Drug: ANEB-001
- Part B - Cohort 5 - Placebo (Placebo Comparator): Subjects receive 30 mg of THC and 1 hour later, 10 mg of ANEB-001
  Interventions: Drug: Placebo
- Part B - Cohort 6 - ANEB-001 (Experimental): Subjects will consume a high fat meal prior to receiving 30 mg of THC and 1 hour later, 10 mg of ANEB-001
  Interventions: Drug: ANEB-001
- Part B - Cohort 6 - Placebo (Placebo Comparator): Subjects will consume a high fat meal prior to receiving 30 mg of THC and 1 hour later, placebo
  Interventions: Drug: Placebo
- Part C - Cohort 7 - ANEB-001 (Experimental): Subjects receive a 40 mg dose of THC and a 10 mg dose of ANEB-001
  Interventions: Drug: ANEB-001
- Part C - Cohort 8 - ANEB-001 (Experimental): Subjects receive a 60 mg dose of THC and a 20 mg dose of ANEB-001
  Interventions: Drug: ANEB-001

INTERVENTIONS:
Drug: ANEB-001 — Experimental Treatment
  Arms: Part A - ANEB-001; Part B - Cohort 1 - ANEB-001; Part B - Cohort 2 - ANEB-001; Part B - Cohort 3 - ANEB-001; Part B - Cohort 4 - ANEB-001; Part B - Cohort 5 - ANEB-001; Part B - Cohort 6 - ANEB-001; Part C - Cohort 7 - ANEB-001; Part C - Cohort 8 - ANEB-001
Drug: Placebo — Placebo comparator
  Arms: Part A - Placebo; Part B - Cohort 1 - Placebo; Part B - Cohort 2 - Placebo; Part B - Cohort 3 - Placebo; Part B - Cohort 4 - Placebo; Part B - Cohort 5 - Placebo; Part B - Cohort 6 - Placebo

SUMMARY:
The aim of this study is to investigate whether ANEB-001 effectively penetrates the brain and inhibits the psychotropic effects of Δ9-Tetrahydrocannabinol (THC), the main psychoactive constituent of cannabis. This randomized, placebo-controlled, double-blind study is designed as a proof-of-pharmacology and dose finding study for the antagonistic effect of ANEB-001 during a THC challenge. Results of this study will inform the future potential use of ANEB-001 as an emergency treatment for acute cannabinoid intoxication.

DETAILED DESCRIPTION:
This study will evaluate whether ANEB-001 effectively inhibits the psychotropic effects of Δ9-Tetrahydrocannabinol (THC). All cohorts in part A and B of the study will be randomized, double-blind and placebo-controlled. Randomization is deemed appropriate to avoid selection bias for active compound or placebo treatment. A double-blind and placebo-controlled design is deemed appropriate because of the safety, tolerability and pharmacodynamic assessments that will be performed in this study. By double-blinding the study, bias arising from study subject's or investigator's knowledge about treatment assignment is avoided. Part C does not include a placebo group and will therefore not be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* BMI between 18 and 30 kg/m2
* Minimum weight 50 kg
* Occasional cannabis user

Exclusion Criteria:

* Evidence of active or chronic condition that could interfere with, or which the treatment of might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator
* Clinically significant abnormalities, as judged by the investigator
* Positive Hepatitis B surface antigen, Hepatitis C antibody or HIV antibody at screening
* Systolic blood pressure greater than 130 or less than 90 mm Hg and diastolic blood pressure greater than 95 or less than 50 mm Hg at screening Abnormal findings in the resting electrocardiogram
* Use of any medications within 7 days of study drug administration, or less than 5 half-lives (whichever is longer). Exceptions are paracetamol and ibuprofen and topical medications.
* Use of any vitamin, mineral, herbal and dietary supplements within 7 days of study drug administration, or less than 5 half-lives (whichever is longer)
* Participation in an investigational drug or device study (last dosing of previous study was within 90 days prior to first dosing of this study)
* History of abuse of addictive substances (alcohol, illegal substances) or current use of more than 21 units alcohol per week, drug abuse, or regular user of sedatives, hypnotics, tranquilizers, or any other addictive agent other than recreative use of THC
* Positive test for drugs of abuse (other than THC) at screening.
* Positive test for drugs of abuse pre-dose
* Clinically significant suicidal ideation in the past 5 years as judged by the investigator or any life-time suicide attempts
* History of cannabis-induced psychosis, schizophrenia or other clinically relevant psychiatric disorders, as judged by the investigator.
* History of a clinically significant mood disorder, including but not limited to major depressive disorder, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-08-26 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Subjective Feeling High | Day 1
  Feeling High on a visual analog scale (mm)
Postural stability | Day 1
  Body sway (mm);
Subjective Alertness | Day 1
  Alertness on a visual analog scale (mm)
Heart Rate | Day 1
  Heart Rate in beats/min

SECONDARY OUTCOMES:
Subjective Mood | Day 1
  Mood on a visual analog scale (mm)
Subjective Calmness | Day 1
  Calmness on a visual analog scale (mm)
Feeling of Drug Effect | Day 1
  Feeling of drug effect on a visual analog scale (mm)
Symbol Digit Substitution Test (SDST) | Day 1
  Part C Only
Visual Verbal Learning Test (VVLT) | Day 1
  Part C Only
Timed Up-and-Go test (TUG) | Day 1
  Part C Only
Alternate Finger Tapping (AFT) | Day 1
  Part C Only
Basic Symptom Inventory (BSI) | Day 1
  Part C Only
Brief Psychiatric Rating Scale (BPRS) | Day 1
  Part C Only
Clinical Global Impression of Severity (CGIS) | Day 1
  Part C Only

CONTACTS AND LOCATIONS:
Overall Officials: GJ Groeneveld, MD, PhD, Principal Investigator — CHDR
Locations (1):
- Centre for Human Drug Research (CHDR), Leiden, South Holland, Netherlands